CLINICAL TRIAL: NCT02427230
Title: The Effect of Pelvic Floor Muscle Training and Neuromuscular Electrical Stimulation on Urinary Incontinence and Quality of Life in Women With Spinal Cord Injury
Brief Title: Treatment of Urinary Incontinence in Women With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Herlev Hospital (Other); University of Copenhagen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Marlene Elmelund, MD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2-2014-113; 20.941 (Other Grant/Funding Number: Gross. L.F. Foghts Fond)
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Spinal Cord Injury; Urinary Incontinence
Keywords: Pelvic Floor Muscle Training; Neuromuscular Electrical Stimulation; Urinary Incontinence; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Incontinence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvic floor muscle training (PFMT) (Active Comparator): Pelvic floor muscle training daily during 12 weeks.
  Interventions: Behavioral: Pelvic floor muscle training
- PFMT and electrical stimulation (Active Comparator): Pelvic floor muscle training and intravaginal neuromuscular electrical stimulation daily during 12 weeks.
  Interventions: Behavioral: Pelvic floor muscle training; Drug: vaginal electrical stimulator (CefarPeristim Pro)

INTERVENTIONS:
Behavioral: Pelvic floor muscle training — The intervention in group 1 consists of three private lessons in PFMT conducted by a physiotherapist every 4th week.
  At each consultation the physiotherapist will use manual palpation of the pelvic floor muscles and Electromyography Biofeedback (EMG). Patients will be instructed to carry out three series of approximately 10 near-maximal pelvic floor muscle contractions held for approximately 6-8 seconds daily during 12 weeks.
  Other Names: Group 1
  Arms: Pelvic floor muscle training (PFMT)
Behavioral: Pelvic floor muscle training — The intervention in group 2 consist of three private lessons in PFMT and intravaginal NMES conducted by a physiotherapist every 4th week.
  At each consultation the physiotherapist will use manual palpation of the pelvic floor muscles and Electromyography Biofeedback (EMG). Patients will be instructed to carry out three series of approximately 10 near-maximal pelvic floor muscle contractions held for approximately 6-8 seconds daily during 12 weeks.
  Additionally, patients will be instructed on how to use intravaginal NMES and each patient receives a vaginal electrical stimulator (CefarPeristim Pro). The NMES settings consist of two different frequencies, 40 Hz and 10 Hz, and patients are instructed to use both settings daily for maximum 30 minutes during 12 weeks.
  Other Names: Group 2
  Arms: PFMT and electrical stimulation
Drug: vaginal electrical stimulator (CefarPeristim Pro) — electrical stimulation
  Arms: PFMT and electrical stimulation

SUMMARY:
The purpose of this study is to determine whether pelvic floor muscle training (PFMT) and intravaginal neuromuscular electrical stimulation (NMES) are effective in reducing urinary incontinence and improving quality of life in women with spinal cord injury (SCI).

DETAILED DESCRIPTION:
SCI patients often experience neurogenic bladder dysfunction with neurogenic detrusor overactivity or areflexic bladder. Due to this, 40-50 % of the SCI population suffers from urinary incontinence, which often reduces the patient's quality of life.

In order to manage the neurogenic bladder dysfunction, SCI patients use specialized bladder emptying methods, most frequently clean intermittent catheterization. To reduce the symptoms of neurogenic detrusor overactivity and urinary incontinence in patients with a SCI, medical anticholinergic therapy can be assessed, but the effect is sparse and many adverse effects have been reported. Injection of Botulinum-A toxin in the bladder has shown great potential in minimizing the symptoms of neurogenic detrusor overactivity and urinary incontinence, though it is an expensive and invasive method that needs to be repeated due to its temporary effect.

PFMT and NMES of the pelvic muscles are non-invasive and cheap treatments without side effects and several studies have demonstrated the positive effect of intravaginal NMES and/or PFMT on urinary incontinence in able-bodied women as well as women with neurological disorders like multiple sclerosis.

Despite the fact that NMES of weak or paralyzed striated muscles has been used for decades in patients suffering from SCI, to our knowledge, no study has previously investigated the effect of PFMT and intravaginal NMES in women with SCI.

The aim of this study is to evaluate the effect of PFMT and intravaginal NMES on Urinary Incontinence and Quality of Life in women with SCI. In particular, we will investigate the potential additional effect of intravaginal NMES, when NMES is conducted in combination with PFMT.

This study is designed as a randomized clinical trial, investigating the effect of PFMT alone and in combination with intravaginal NMES. We will include 40 female patients with an incomplete SCI and urinary incontinence. After physiotherapeutic guidance, the patients perform PFMT or PFMT + NMES daily at home for 12 weeks with follow-up evaluations every fourth week.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete SCI graded C, D og E on ASIA Impairment Scale, sustained minimum 3 months ago
* urinary incontinence, corresponding to a total ICIQ-UI-SF score ≥ 8

Exclusion Criteria:

* Regular treatment with botox bladder injections or < 1 year since last botox injection
* Lack of urodynamic investigation after the SCI
* Pregnancy
* Pacemaker
* Lack of ability to contract the pelvic floor muscles during objective clinical examination

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire, Urinary Incontinence, Short Form (ICIQ-UI-SF) | up to week 24

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire, Overactive Bladder (ICIQ-AOB) | up to week 24
Urethral Pressure Reflectometry (UPR) parameters | up to week 24
  UPR is a novel method of measuring the pressure and cross-sectional area in the female urethra
3 days voiding diary | 3 days
24 hour pad test | 24 hour
International Spinal Cord Injury Quality of Life Basic Data Set | up to week 24
Patient Global Index of Improvement scale (PGI-I) | up to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Elmelund, MD, Principal Investigator — Clinic for Spinal Cord Injuries, Glostrup University Hospital/Rigshospitalet and Department of Gynaecology and Obstetrics, Herlev University Hospital; Fin Biering-Sørensen, MD DMSc Prof, Study Director — Clinic for Spinal Cord Injuries, Glostrup University Hospital/Rigshospitalet; Niels Klarskov, MD Lecturer, Study Director — Department of Gynaecology and Obstetrics, Herlev University Hospital
Locations (1):
- Department of Gynaecology and Obstetrics, Herlev University Hospital, Herlev, Denmark

REFERENCES:
- [Background] Hansen RB, Biering-Sorensen F, Kristensen JK. Urinary incontinence in spinal cord injured individuals 10-45 years after injury. Spinal Cord. 2010 Jan;48(1):27-33. doi: 10.1038/sc.2009.46. Epub 2009 Jun 2. PMID 19488052
- [Background] Jerez-Roig J, Souza DL, Espelt A, Costa-Marin M, Belda-Molina AM. Pelvic floor electrostimulation in women with urinary incontinence and/or overactive bladder syndrome: a systematic review. Actas Urol Esp. 2013 Jul-Aug;37(7):429-44. doi: 10.1016/j.acuro.2012.08.003. Epub 2012 Dec 13. English, Spanish. PMID 23246103
- [Background] McClurg D, Ashe RG, Marshall K, Lowe-Strong AS. Comparison of pelvic floor muscle training, electromyography biofeedback, and neuromuscular electrical stimulation for bladder dysfunction in people with multiple sclerosis: a randomized pilot study. Neurourol Urodyn. 2006;25(4):337-48. doi: 10.1002/nau.20209. PMID 16637070
- [Background] McClurg D, Ashe RG, Lowe-Strong AS. Neuromuscular electrical stimulation and the treatment of lower urinary tract dysfunction in multiple sclerosis--a double blind, placebo controlled, randomised clinical trial. Neurourol Urodyn. 2008;27(3):231-7. doi: 10.1002/nau.20486. PMID 17705160
- [Background] Bo K, Talseth T, Holme I. Single blind, randomised controlled trial of pelvic floor exercises, electrical stimulation, vaginal cones, and no treatment in management of genuine stress incontinence in women. BMJ. 1999 Feb 20;318(7182):487-93. doi: 10.1136/bmj.318.7182.487. PMID 10024253
- [Background] Klarskov N, Lose G. Urethral pressure reflectometry; a novel technique for simultaneous recording of pressure and cross-sectional area in the female urethra. Neurourol Urodyn. 2007;26(2):254-61. doi: 10.1002/nau.20283. PMID 17016844